CLINICAL TRIAL: NCT01575548
Title: Randomized, Double-Blind Phase III Study of Pazopanib vs. Placebo in Patients With Metastatic Renal Cell Carcinoma Who Have No Evidence of Disease Following Metastatectomy
Brief Title: Pazopanib Hydrochloride in Treating Patients With Metastatic Kidney Cancer Who Have No Evidence of Disease After Surgery
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-00723; NCI-2012-00723 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000730383; ECOG-E2810; E2810; E2810 (Other: ECOG-ACRIN Cancer Research Group); E2810 (Other: CTEP); U10CA021115 (NIH); U10CA180820 (NIH); U10CA180830 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2012-04-10; First posted 2012-04-11 (Estimated); Results first posted 2022-07-19 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Clear Cell Renal Cell Carcinoma; Stage IV Renal Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Magnetic Resonance Spectroscopy; pazopanib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Pazopanib) (Experimental): Patients receive pazopanib hydrochloride PO QD on days 1-28. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI throughout the study.
  Interventions: Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Pazopanib Hydrochloride; Other: Questionnaire Administration
- Arm B (Placebo) (Placebo Comparator): Patients receive placebo PO QD on days 1-28. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI throughout the study.
  Interventions: Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Pazopanib Hydrochloride — Given PO
  Other Names: GW 786034B; GW-786034B; GW786034B; Pazopater; Votrient
  Arms: Arm A (Pazopanib)
Other: Placebo Administration — Given PO
  Arms: Arm B (Placebo)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase III trial studies how well pazopanib hydrochloride works compared to placebo in treating patients with kidney cancer that has spread to other parts of the body and have no evidence of disease after surgery. Pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate disease-free survival with pazopanib (pazopanib hydrochloride) as compared to placebo, defined as the time from randomization to the development of recurrent disease, second primary cancer (other than localized breast, localized prostate, or non-melanoma skin cancer) or death from any cause for patients with metastatic renal cell carcinoma (RCC) with no evidence of disease following metastasectomy.

SECONDARY OBJECTIVES:

I. To describe the overall survival of patients with advanced RCC randomly assigned to receive placebo or pazopanib for one year following metastasectomy to no evidence of disease (NED).

II. To describe treatment and (at recurrence) disease-related adverse events in the two treatment arms.

III. To analyze quality-adjusted time without symptoms of disease or treatment (Q-TWiST) for subjects in the two treatment arms.

IV. To characterize changes in patient-reported fatigue and (at recurrence) kidney cancer-related symptoms during and following treatment with pazopanib compared to placebo.

V. To explore the association between plasma trough levels of pazopanib and disease-free and overall survival.

VI. To prospectively bank preserved tissue from primary tumors and associated metastatic sites in patients with RCC.

OUTLINE: Patients are randomized to 1of 2 treatment arms.

ARM A: Patients receive pazopanib hydrochloride orally (PO) once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive placebo PO QD on days 1-28. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.

Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) throughout the study.

After completion of study treatment, patients are followed up every 3 months for the first two years, every 6 months for the next 3 years, and then annually up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years of age at the time of randomization
* Patient must have pathologically confirmed renal cell carcinoma with a clear cell component; pure papillary and chromophobe histologies are excluded; there must be pathologic confirmation of metastatic disease in the resected metastasectomy specimen
* Patient must have undergone nephrectomy or partial nephrectomy to remove primary renal cell carcinoma (at any time in the past)
* Patient must have undergone surgical resection to remove one or more sites of metastatic disease, with successful removal of all known sites 2-12 weeks prior to randomization. Any number of prior metastasectomies may have been performed in the past, so long as the most recent procedure was within the 12 weeks of registration. The most recent procedure may be nephrectomy for a renal primary tumor
* Patients with synchronous disease at initial diagnosis must have metastatic (M1) disease (American Joint Committee on Cancer [AJCC] 7th edition T1-4N0-1M1)
* Positive surgical margins are permitted if the surgeon confirms complete resection of gross metastatic disease, and post-operative scans are negative
* Patients presenting with metachronous disease may have distant metastases, regional lymph node or renal bed recurrence. Recurrences at a partial nephrectomy resection site are not eligible if it is the only site of disease
* Patient must have no evidence of disease on post-operative imaging:

  * A computed tomography (CT) of the chest must be obtained within 4 weeks prior to randomization with or without contrast
  * A CT of the abdomen/pelvis must be obtained within 4 weeks prior to randomization with intravenous (IV) contrast (oral contrast may be added at the radiologist's discretion); an magnetic resonance imaging (MRI) of the abdomen/pelvis with gadolinium may be substituted for the CT if the CT with IV contrast is contra-indicated
  * An MRI of the brain with and without gadolinium must be done within 8 weeks prior to randomization; a CT of the brain with and without IV contrast is permitted if MRI is contra-indicated (i.e., pacemaker)
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at the time of randomization
* Absolute granulocyte count > 1,500/mcL (within 2 weeks prior to randomization)
* Platelets > 100,000/mcL (within 2 weeks prior to randomization)
* Total bilirubin < 1.5 x institutional upper limit of normal (ULN) (within 2 weeks prior to randomization)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 x upper limit of normal (ULN) (within 2 weeks prior to randomization)
* Calculated creatinine clearance (CrCl) > 30 mL/min (within 2 weeks prior to randomization)
* Subjects must have a urine protein/creatinine (UPC) ratio < 1; if UPC >= 1, then a 24-hour urine total protein must be obtained; subjects must have a 24-hour urine protein value < 1 g to be eligible; use of urine dipstick for renal function assessment is not acceptable (within 2 weeks prior to randomization)
* All females of childbearing potential must have a blood test or urine study within 2 weeks prior to randomization to rule out pregnancy; a female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method of contraception or to abstain from sexual intercourse for the duration of their participation in the study; should a woman become pregnant while participating in this study, she should inform her treating physician immediately; if a man impregnates a woman while participating in this study, he should inform his treating physician immediately
* Patient must be able to swallow pills and have no significant impairment in gastrointestinal absorption including history of gastric bypass surgery
* Patient must have a corrected QT (QTc) interval on electrocardiogram (ECG) =< 0.48 seconds by Bazett's calculation (=< Common Terminology Criteria for Adverse Events [CTCAE] version [v.]4 grade 2) prior to randomization
* Patient must have a systolic blood pressure =< 140 mmHg and diastolic blood pressure must be =< 90 mmHg, measured within 4 weeks prior to randomization; initiation or adjustment of anti-hypertensives prior to starting study treatment is allowed
* Patient must have no history of cerebrovascular accident (CVA) within 6 months of randomization

Exclusion Criteria:

* Patients presenting with tumors within the kidneys (multiple synchronous or single/multiple metachronous) are not eligible if there are no extrarenal sites of disease (i.e. potential multifocal primary disease)
* Patient must not have received any prior or concurrent systemic therapy for RCC. Adjuvant placebo administration is permitted
* Patient must have no active peptic ulcer disease
* Patient must have no active inflammatory bowel disease
* Patient must have no New York Heart Association (NYHA) class II or greater congestive heart failure
* Patient must have no prior history or current clinically apparent central nervous system metastases
* Women must not be pregnant or breast-feeding due to the unknown effects of pazopanib on the developing fetus
* Patient must have no history of allergic reactions attributed to compounds of similar chemical or biologic composition to pazopanib
* Patient must have no uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patient must not have serious or non-healing wound, ulcer, or bone fracture at the time of randomization
* Patient must have no history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 4 weeks prior to randomization
* Patient must have no history of myocardial infarction, hospital admission for unstable angina, cardiac angioplasty or stenting within 6 months of randomization
* Patient must have no history venous thrombosis within 12 weeks of randomization
* Patient cannot be taking strong cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors such as:

  * Antibiotics: clarithromycin, telithromycin, troleandomycin
  * Human immunodeficiency virus (HIV) antiviral protease inhibitors: ritonavir, indinavir, saquinavir, nelfinavir, amprenavir, lopinavir
  * Antifungals: itraconazole, ketoconazole, voriconazole, fluconazole
  * Antidepressants: nefazodone
* Patient must not have history of hemoptysis in excess of 2.5 mL (1/2 teaspoon) within 8 weeks prior to randomization
* Patient must not be taking drugs known to prolong the QTc interval; such drugs should be discontinued at least 5 half-lives prior to randomization
* Patients must not have any history of other cancer within 3 years from time of randomization with the exception of basal cell skin cancer, squamous cell skin cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast, or resected non-invasive (Ta) urothelial carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2012-08-08 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2026-02-21 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard J Appleman, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (581):
- United States (581):
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - PCR Oncology, Arroyo Grande, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Newman Regional Health, Emporia, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - East Jefferson General Hospital, Metairie, Louisiana
  - Robert Veith MD LLC, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - William Beaumont Hospital-Grosse Pointe, Grosse Pointe, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Monroe Cancer Center, Monroe, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - Michigan Cancer Specialists, Roseville, Michigan
  - Oakland Colon Rectal Associates, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Hematology Oncology Consultants PC-Royal Oak, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Premier Hematology Oncology Care, Sterling Heights, Michigan
  - Mitchell Folbe MD PC, Sterling Heights, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Claudia BR Herke MD PC, Troy, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Garnet Health Medical Center, Middletown, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Randolph Hospital, Asheboro, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Sampson Radiation Oncology, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Trinity's Tony Teramana Cancer Center, Steubenville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - Cancer Care Associates-Norman, Norman, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Integris Cancer Institute of Oklahoma, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Warren Clinic Oncology-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - Providence Medford Medical Center, Medford, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Roper Hospital, Charleston, South Carolina
  - Charleston Oncology - Roper, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-North Charleston, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Charleston, South Carolina
  - Charleston Oncology - Saint Francis, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-West Ashley, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Lowcountry Hematology Oncology PA-Mount Pleasant, Mt. Pleasant, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Bristol, Bristol, Tennessee
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Farmington Health Center, Farmington, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Ballad Health Cancer Care - Bristol, Bristol, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Medical Center, Bellevue, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Lakeview Medical Center-Marshfield Clinic, Rice Lake, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Appleman LJ, Kim SE, Harris WB, Pal SK, Pins MR, Kolesar J, Agarwal N, Parikh RA, Vaena DA, Ryan CW, Hashmi M, Costello BA, Cella D, Dutcher JP, DiPaola RS, Haas NB, Wagner LI, Carducci MA. Randomized, Double-Blind Phase III Study of Pazopanib Versus Placebo in Patients With Metastatic Renal Cell Carcinoma Who Have No Evidence of Disease After Metastasectomy: ECOG-ACRIN E2810. J Clin Oncol. 2024 Jun 10;42(17):2061-2070. doi: 10.1200/JCO.23.01544. Epub 2024 Mar 26. PMID 38531002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on August 8, 2012 and closed to accrual on July 25, 2017, with a total enrollment of 129 patients.
Groups:
- Arm A (Pazopanib): Patients receive pazopanib hydrochloride PO QD on days 1-28. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.
- Arm B (Placebo): Patients receive placebo PO QD on days 1-28. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm A (Pazopanib) | Arm B (Placebo)
Started | 66 | 63
Received Protocol Therapy | 63 | 61
Completed | 26 | 30
Not Completed | 40 | 33
Not completed — Adverse Event | 15 | 2
Not completed — Disease progression | 12 | 25
Not completed — Death | 1 | 0
Not completed — Other complicating disease | 1 | 0
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Noncompliance | 1 | 0
Not completed — Anticipated surgery | 0 | 1
Not completed — Never started protocol therapy | 3 | 2

BASELINE CHARACTERISTICS:
Population: All randomized patients are included in this analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Pazopanib) | Arm B (Placebo) | Total
Number analyzed (Participants) | 66 | 63 | 129
Age, Continuous [Median (Full Range); unit: years] | 60 [40 to 85] | 61 [31 to 80] | 60 [31 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 27 | 48
  Male | 45 | 36 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 60 | 61 | 121
  Unknown or Not Reported | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 61 | 57 | 118
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS)
Description: Disease-free survival (DFS) is defined as the time from randomization to the development of recurrent disease, second primary cancer (other than localized breast, localized prostate, or non-melanoma skin cancer) or death from any cause.
Time Frame: Assessed every 3 months for the first 2 years, every 6 months for the next 3 years, and then annually up to 6 years
Population: All randomized patients are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Pazopanib) | Arm B (Placebo)
Number analyzed (Participants) | 66 | 63
months | 17 [14.0 to 20.4] | 14.2 [9.1 to 23.5]
Statistical Analysis 1: Comparison: Arm A (Pazopanib) vs Arm B (Placebo); Test type: Superiority; p = 0.21, Log Rank; Stratified log rank test was used to compare DFS between the two arms; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.54 to 1.29]

2. Secondary Outcome: 3-year Overall Survival (OS) Rate
Description: Overall survival is defined as the time from randomization to death or date last known alive. Kaplan-Meier method was used to estimate 3-year overall survival rate.
Time Frame: Assessed every 3 months for the first 2 years, and then every 6 months for the 3rd year.
Population: All randomized patients are included in this analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Pazopanib) | Arm B (Placebo)
Number analyzed (Participants) | 66 | 63
proportion of participants | 0.816 [0.712 to 0.935] | 0.889 [0.798 to 0.990]

3. Secondary Outcome: Quality-adjusted Time Without Symptoms of Disease or Treatment (Q-TWiST)
Description: OS for each arm is divided into 3 health states: toxicity (TOX), time without symptoms of disease or toxicity (TWiST), and recurrence (REC). TOX is defined as the time spent with grade 3/4 adverse events (AEs) prior to disease recurrence. TWiST is defined as the time prior to disease recurrence when no AEs of grade 3/4 were experienced. REC health state is defined as the time from disease recurrence or second primary cancer until death. Patients alive will be censored at the date of last contact. For each health state, a patient-reported utility weight will be assigned. The mean amount of time in each state will be estimated using Kaplan and Meier method.
  TWiST = mean recurrence-free survival (RFS) - mean time with toxicities REC = mean OS - mean RFS Q-TWiST = (uTOX x TOX) + (uTWiST x TWiST) + (uREC x REC) Where uTOX, uTWiST, and uREC represent the average group utility value for each state for that arm and TOX, TWiST and REC represent the mean duration of the state for that arm.
Time Frame: Assessed every 3 months for the first 2 years, every 6 months for the next 3 years, then annually up to 10 years
Reporting Status: Not Posted, anticipated posting 2026-12

4. Secondary Outcome: Change in Functional Assessment of Chronic Illness Therapy (FACIT) - Fatigue Score From Baseline to 6 Months
Description: FACIT-Fatigue subscale (13 items) was used to evaluate fatigue in this patient population. The score ranges between 0 and 52. The higher the score, the better the quality of life. The change in FACIT-Fatigue score from baseline to 6 months will be compared between the two arms.
Time Frame: Assessed at baseline and 6 months
Reporting Status: Not Posted, anticipated posting 2026-12

5. Secondary Outcome: Change in Functional Assessment of Cancer Therapy-Kidney Symptom Index Score From Baseline to 6 Months
Description: Functional Assessment of Cancer Therapy Kidney Cancer Symptom Index - 15 Item Version (FKSI-15) will be used to evaluate the quality of life concerns among this patient population. The change in score from baseline to 6 months will be compared between the two arms. The score ranges between 0 and 60. A score of "0" is a severely symptomatic patient and the highest possible score is an asymptomatic patient.
Time Frame: Assessed at baseline and 6 months
Reporting Status: Not Posted, anticipated posting 2026-12

6. Secondary Outcome: Change in Plasma Levels of Pazopanib From Baseline to Cycle 2 Day 1
Description: Plasma concentration of pazopanib will be assessed at baseline and cycle 2 day 1.
Time Frame: Assessed at baseline and cycle 2 day 1
Reporting Status: Not Posted, anticipated posting 2026-12

7. Other Pre Specified Outcome: To Prospectively Bank Preserved Tissue From Primary Tumors and Associated Metastatic Sites in Patients With RCC
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment
Description: Serious adverse events (SAEs) are defined as AEs of grade 3 or higher that are possibly, probably, or definitely related to protocol treatment. Other AEs are defined as those adverse events of grade 1 or grade 2 that are possibly, probably, or definitely related to protocol treatment with a frequency of at least 5% in a given arm.
  All randomized patients were included in the all-cause mortality table. Only patients who received assigned treatment were included in the SAE and other AE tables.
Arm/Group | Arm A (Pazopanib) | Arm B (Placebo)
All-Cause Mortality (participants affected / at risk) | 15/66 | 6/63
Serious Adverse Events (participants affected / at risk) | 43/63 | 14/61
Other Adverse Events (participants affected / at risk) | 62/63 | 49/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Pazopanib) (N=63) | Arm B (Placebo) (N=61)
Fatigue (General disorders) | 3 | 1
General disorders and administration site conditions - Other (General disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 10 | 0
Jejunal hemorrhage (Gastrointestinal disorders) | 1 | 0
Jejunal ulcer (Gastrointestinal disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Bronchial infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 9 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 0
Lipase increased (Investigations) | 4 | 2
Lymphocyte count decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 0
Serum amylase increased (Investigations) | 1 | 0
Weight loss (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 0 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 2 | 0
Hypertension (Vascular disorders) | 20 | 4
Thromboembolic event (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Pazopanib) (N=63) | Arm B (Placebo) (N=61)
Fatigue (General disorders) | 39 | 20
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 | 4
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 7 | 0
Abdominal pain (Gastrointestinal disorders) | 14 | 6
Diarrhea (Gastrointestinal disorders) | 41 | 14
Nausea (Gastrointestinal disorders) | 37 | 15
Vomiting (Gastrointestinal disorders) | 18 | 2
Alanine aminotransferase increased (Investigations) | 24 | 8
Aspartate aminotransferase increased (Investigations) | 20 | 7
Blood bilirubin increased (Investigations) | 7 | 0
Lymphocyte count decreased (Investigations) | 12 | 2
Neutrophil count decreased (Investigations) | 12 | 1
Platelet count decreased (Investigations) | 25 | 4
White blood cell decreased (Investigations) | 19 | 1
Anorexia (Metabolism and nutrition disorders) | 15 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 11 | 11
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 10 | 4
Dizziness (Nervous system disorders) | 6 | 10
Headache (Nervous system disorders) | 28 | 12
Proteinuria (Renal and urinary disorders) | 14 | 10
Hypertension (Vascular disorders) | 41 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT01575548/Prot_SAP_001.pdf